CLINICAL TRIAL: NCT06672328
Title: Action Observation Training for Functional Performance in Children with Cerebral Palsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/40
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Cerebral Palsy (CP); Physical Functional Performance
Keywords: Balance; Cerebral Palsy; Physical Function Performance; Mobility; Spasticity
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional Group (Experimental): The participants will receive AOT based mobility and balance exercises along with conventional therapy consisting of simple lower limb stretchings and strengthening .
  The AOT-based exercises include different exercises in sitting, standing and turning stances.
  The fun based activities inlcude reaching for objects, tower building and taking turns in various stances.
  Interventions: Procedure: Training with Action Observation Therapy
- Control Group (Active Comparator): The participants will receive mobility and balance exercises without Action Obseravtion along with conventional therapy consisting of simple lower limb stretchings and strengthening .
  The AOT-based exercises include different exercises in sitting, standing and turning stances.
  The fun based activities inlcude reaching for objects, tower building and taking turns in various stances.
  Interventions: Procedure: Training without Action Observation Therapy

INTERVENTIONS:
Procedure: Training with Action Observation Therapy — AOT based mobility and balance exercises along with conventional therapy consisting of simple lower limb stretchings and strengthening.
  The fun based activities inlcude reaching for objects, tower building and taking turns in various stances.
  Arms: Interventional Group
Procedure: Training without Action Observation Therapy — Cerebral Palsy patients will receive balance and mobility training without action observation in various stances of sitting, standing and turning.
  Activities are fun based and include reaching for objects, tower building and taking turns in different positions.
  Arms: Control Group

SUMMARY:
This study is a randomized control trial and aims to determine the effects of Action Observation on balance and mobility in patients with cerebral palsy compared to training without action observation.

DETAILED DESCRIPTION:
Effetcs of Action observation will be assessed for functional performance which includes the parameters of balance and mobility.

Spastic CP children agd 5-12 will be recruited in the study. The participants would be assessed through Modified Ashworth scale, GMFCS, Pediatrics balance scale and GMFM-88 .

Informed Consent will ne taken after which the participants will be recruited into the two groups, where one group will recieve training with Action observation and other group will receive training without Action observation.

Baseline and Post-treatment measurements will be taken for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-12.
* Spastic CP.
* Modified Ashworth Scale spasticity score 0-2
* GMFCS level I, II or III.
* Able to understand and follow commands, e.g. "Stand up, please".
* Able to sit to stand with or without assistance.

Exclusion Criteria:

* Any orthopedic procedure in the past 6 months, that could prevent exercise training.
* Any co-morbid condition such as spinal atrophy, osteogenesis imperfecta etc.
* History of chronic seizure attacks.
* Children with severe visual/hearing impairments.
* Presence of knee contractures

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-09-10 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Static balance | 8 weeks
  Pediatrics berg balance scale will be used for balance assessment. It has a total score of 56, with higher scores indicating better balance.
Dynamic balance | 8 weeks
  Pediatrics berg balance scale will be used for balance assessment. It has a total score of 56, with higher scores indicating better balance
Mobility | 8 weeks
  GMFM-88 scale will be used for assessment of mobility, particularly the subscales B,D and E related to mobility in sitting, standing and walking stances.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Thrapy, Islamabad, Pakistan